CLINICAL TRIAL: NCT00611884
Title: A 16 Week Randomised, Open-labelled, Four-armed, Treat-to-target, Parallel-group Trial Comparing SIBA D Once Daily, SIBA E Once Daily, SIBA D Monday, Wednesday and Friday and Insulin Glargine Once Daily, All in Combination With Metformin in Subjects With Type 2 Diabetes Failing on OAD Treatment
Brief Title: Comparison of Two NN1250 Formulations Versus Insulin Glargine, All in Combination With Metformin in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1250-1836
Record Dates: First submitted 2008-01-29; First posted 2008-02-11 (Estimated); Results first posted 2015-11-16 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; insulin degludec; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- SIBA (D) (Experimental)
  Interventions: Drug: insulin degludec; Drug: metformin
- SIBA (E) (Experimental)
  Interventions: Drug: insulin degludec; Drug: metformin
- SIBA (D) M, W, F (Experimental)
  Interventions: Drug: insulin degludec; Drug: metformin
- IGlar (Active Comparator)
  Interventions: Drug: insulin glargine; Drug: metformin

INTERVENTIONS:
Drug: insulin glargine — Treat-to-target dose titration scheme, s.c. injection.
  Arms: IGlar
Drug: insulin degludec — Formulation D: Treat-to-target dose titration scheme, s.c. injection, once daily
  Arms: SIBA (D)
Drug: insulin degludec — Formulation E: Treat-to-target dose titration scheme, s.c. injection, once daily
  Arms: SIBA (E)
Drug: insulin degludec — Formulation D: Treat-to-target dose titration scheme, s.c. injection, 3 times weekly
  Arms: SIBA (D) M, W, F
Drug: metformin — Tablets, 1500-2000 mg/day

SUMMARY:
This trial is conducted in Africa, Asia and North America. The aim of this trial is to compare two insulin degludec (NN1250, SIBA) formulations with each other and with insulin glargine, all in combination with metformin in insulin naive subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. (Trial-related activities are any procedure that would not have been performed during normal management of the subject.)
* Insulin naïve type 2 diabetes subjects (as diagnosed clinically) for at least 3 months (no previous insulin treatment or previous short term insulin treatment maximeum 14 days within the last 3 months)
* Treatment with one or two oral anti-diabetic drug (OADs): metformin, sulphonylurea (SU) (or other insulin secretagogue e.g. repaglinide, nateglinide), alpha-glucosidase inhibitors for at least 2 months at a stable maximally tolerated dose or at least half maximally allowed dose according to the summary of product characteristics (SPC) or locally approved PI
* HbA1c 7.0-11.0 % (both inclusive)
* Body Mass Index (BMI) 23-42 kg/m^2 [lb/in^2 x 703] (both inclusive)

Exclusion Criteria:

* Metformin contraindication according to local practice
* Thiazolidinedione (TZD) treatment within previous three months prior to visit 1
* Any systemic treatment with products which in the Investigator's opinion could interfere with glucose or lipid metabolism (e.g. systemic corticosteroids) three months prior to randomisation
* Subject has a clinically significant, active (during the past 12 months) disease of the gastrointestinal, pulmonary, neurological, genitourinary, or haematological system (except for conditions associated with type 2 diabetes) that, in the opinion of the Investigator, may confound the results of the trial or pose additional risk in administering trial drug

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2008-01; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (26):
- United States (17):
  - Novo Nordisk Investigational Site, Inglewood, California
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Redlands, California
  - Novo Nordisk Investigational Site, Spring Valley, California
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Idaho Falls, Idaho
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Springfield, Illinois
  - Novo Nordisk Investigational Site, Greensboro, North Carolina
  - Novo Nordisk Investigational Site, Medford, Oregon
  - Novo Nordisk Investigational Site, Simpsonville, South Carolina
  - Novo Nordisk Investigational Site, Kingsport, Tennessee
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Newport News, Virginia
  - Novo Nordisk Investigational Site, Renton, Washington
  - Novo Nordisk Investigational Site, Milwaukee, Wisconsin
- Canada (3):
  - Novo Nordisk Investigational Site, Cambridge, Ontario
  - Novo Nordisk Investigational Site, Etobicoke, Ontario
  - Novo Nordisk Investigational Site, Toronto, Ontario
- India (4):
  - Novo Nordisk Investigational Site, Hyderabad, Andhra Pradesh
  - Novo Nordisk Investigational Site, Kochi, Kerala
  - Novo Nordisk Investigational Site, Mumbai, Maharashtra
  - Novo Nordisk Investigational Site, Vellore, Tamil Nadu
- South Africa (2):
  - Novo Nordisk Investigational Site, Johannesburg, Gauteng
  - Novo Nordisk Investigational Site, Durban, KwaZulu-Natal

REFERENCES:
- [Result] Zinman B, Fulcher G, Rao PV, Thomas N, Endahl LA, Johansen T, Lindh R, Lewin A, Rosenstock J, Pinget M, Mathieu C. Insulin degludec, an ultra-long-acting basal insulin, once a day or three times a week versus insulin glargine once a day in patients with type 2 diabetes: a 16-week, randomised, open-label, phase 2 trial. Lancet. 2011 Mar 12;377(9769):924-31. doi: 10.1016/S0140-6736(10)62305-7. PMID 21396703
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 28 sites: Canada (4), India (4), South Africa (3) and the United States of America (17).
Pre-assignment Details: Subjects underwent a run-in period of 3 weeks; 2 weeks of up-titration period, where metformin was up-titrated to 1500 or 2000 mg/day, followed by 1 week of maintenance period. Subjects who tolerated 1500 or 2000 mg/day of metformin for a week and had a median fasting plasma glucose ≥ 7.5 mmol/L (135 mg/dL) were randomised.
Groups:
- SIBA (D): Soluble Insulin Basal Analogue D (SIBA D, 900 nmol/mL [1 dosing unit = 9 nmol], insulin degludec; formulation D) was given subcutaneously once daily (OD) in the evening in combination with at least 1500 mg/day metformin (tablets) for 16 weeks. Insulin doses were initiated at 10 units (U)/day and individually adjusted.
- SIBA (E): Soluble Insulin Basal Analogue E (SIBA E, 600 nmol/mL (1 dosing unit = 6 nmol), insulin degludec; formulation E) was given subcutaneously once daily (OD) in the evening in combination with at least 1500 mg/day metformin (tablets) for 16 weeks. Insulin doses were initiated at 10 U/day and individually adjusted.
- SIBA (D) M, W, F: Soluble Insulin Basal Analogue D (SIBA D, 900 nmol/mL (1 dosing unit = 9 nmol), insulin degludec; formulation D) was given subcutaneously thrice weekly (Monday [M], Wednesday[W], Friday[F]) in the evening in combination with at least 1500 mg/day metformin (tablets) for 16 weeks. Insulin doses were were initiated at 20 U/day and individually adjusted.
- IGlar: Insulin glargine (IGlar) was given subcutaneously once daily (OD) before bedtime in combination with at least 1500 mg/day metformin (tablets) for 16 weeks. Insulin doses were initiated at 10 U/day and individually adjusted.
Period: Overall Study
Arm/Group | SIBA (D) | SIBA (E) | SIBA (D) M, W, F | IGlar
Started | 61 | 60 | 62 | 62
Exposed | 58 (Three subjects withdrew prior to exposure to trial drug) | 59 (One subject withdrew prior to exposure to trial drug) | 61 (One subject withdrew prior to exposure to trial drug) | 61 (One subject withdrew prior to exposure to trial drug)
Completed | 52 | 51 | 58 | 56
Not Completed | 9 | 9 | 4 | 6
Not completed — Adverse Event | 1 | 0 | 0 | 1
Not completed — Non-Compliance | 1 | 4 | 2 | 2
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0
Not completed — Unclassified | 7 | 4 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SIBA (D) | SIBA (E) | SIBA (D) M, W, F | IGlar | Total
Number analyzed (Participants) | 61 | 60 | 62 | 62 | 245
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (8.5) | 55.3 (8.7) | 54.4 (8.8) | 53.1 (10.2) | 54.2 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 27 | 34 | 25 | 108
  Male | 39 | 33 | 28 | 37 | 137
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 8.7 (1.1) | 8.6 (1.2) | 8.8 (1.1) | 8.7 (1.1) | 8.7 (1.1)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] | 10.6 (3.6) | 9.9 (3.2) | 10.6 (3.4) | 9.8 (3.1) | 10.2 (3.4)

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Haemoglobin (HbA1c)
Description: Change from baseline in HbA1c after 16 weeks of treatment
Time Frame: Week 0, Week 16
Population: The full analysis set (FAS) included all randomised subjects and missing data is imputed using last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | SIBA (D) | SIBA (E) | SIBA (D) M, W, F | IGlar
Number analyzed (Participants) | 61 | 60 | 62 | 62
percentage of glycosylated haemoglobin | -1.26 (1.11) | -1.28 (1.11) | -1.46 (1.06) | -1.49 (1.12)

2. Secondary Outcome: Mean of 9-point Self Measured Plasma Glucose Profile (SMPG)
Description: Mean of SMPG after 16 weeks of treatment. Plasma glucose measured: before breakfast, 120 minutes after start of breakfast, before lunch, 120 minutes after start of lunch, before dinner, 120 minutes after start of dinner, before bedtime, at 4 am and before breakfast.
Time Frame: Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | SIBA (D) | SIBA (E) | SIBA (D) M, W, F | IGlar
Number analyzed (Participants) | 61 | 60 | 62 | 62
mmol/L | 8.30 (0.42) | 8.55 (0.42) | 8.45 (0.42) | 8.42 (0.41)

3. Secondary Outcome: Rate of Major and Minor Hypoglycaemic Episodes
Description: Rate of major and minor hypoglycaemic episodes per 100 patient years of exposure (PYE). Major if unable to treat her/himself. Minor if able to treat her/himself and plasma glucose below 3.1 mmol/L.
Time Frame: Week 0 to Week 16 + 5 days follow up
Population: The full analysis set (FAS) included all randomised subjects.
Measure: Number; unit: Episodes/100 years of patient exposure
Arm/Group | SIBA (D) | SIBA (E) | SIBA (D) M, W, F | IGlar
Number analyzed (Participants) | 61 | 60 | 62 | 62
Episodes/100 years of patient exposure
  Major | 0 | 0 | 6 | 0
  Minor | 89 | 60 | 221 | 113

4. Secondary Outcome: Rate of Nocturnal Major and Minor Hypoglycaemic Episodes
Description: Rate of nocturnal major and minor hypoglycaemic episodes per 100 patient years of exposure (PYE). Major if unable to treat her/himself. Minor if able to treat her/himself and plasma glucose below 3.1 mmol/L. Episodes were defined as nocturnal if the time of onset was between 23:00 (included) and 05:59 (included).
Time Frame: Week 0 to Week 16 + 5 days follow up
Population: The full analysis set (FAS) included all randomised subjects.
Measure: Number; unit: Episodes/100 years of patient exposure
Arm/Group | SIBA (D) | SIBA (E) | SIBA (D) M, W, F | IGlar
Number analyzed (Participants) | 61 | 60 | 62 | 62
Episodes/100 years of patient exposure
  Major | 0 | 0 | 6 | 0
  Minor | 6 | 12 | 17 | 0

5. Secondary Outcome: Rate of Treatment Emergent Adverse Events (AEs)
Description: Corresponds to rate of AEs per 100 patient years of exposure. Severity assessed by investigator. Mild: no or transient symptoms, no interference with subject's daily activities. Moderate: marked symptoms, moderate interference with subject's daily activities. Severe: considerable interference with subject's daily activities, unacceptable. Serious AE: AE that at any dose results in any of the following: death, a life-threatening experience, in-subject hospitalization/prolongation of existing hospitalisation, persistent/significant disability/incapacity/congenital anomaly/birth defect.
Time Frame: Week 0 to Week 16 + 5 days follow up
Population: The safety analysis set included all subjects who received at least one dose of the investigational product or its comparator.
Measure: Number; unit: Events/100 years of patient exposure
Arm/Group | SIBA (D) | SIBA (E) | SIBA (D) M, W, F | IGlar
Number analyzed (Participants) | 57 | 59 | 62 | 61
Events/100 years of patient exposure
  Adverse events (AEs) | 594 | 430 | 488 | 622
  Serious AEs | 6 | 0 | 5 | 0
  Severe AEs | 12 | 6 | 0 | 28
  Moderate AEs | 114 | 102 | 110 | 141
  Mild AEs | 468 | 323 | 379 | 452
  Fatal | 0 | 0 | 0 | 0

6. Secondary Outcome: Laboratory Safety Parameters (Biochemistry): Alanine Aminotransferase (ALAT)
Description: Mean values at Week -4 and at Week 16
Time Frame: Week -4, Week 16
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | SIBA (D) | SIBA (E) | SIBA (D) M, W, F | IGlar
Number analyzed (Participants) | 57 | 59 | 62 | 61
IU/L
  ALAT, Week -4, N=56, 59, 62, 60 | 34.6 (19.9) | 29.2 (16.3) | 30.9 (16.0) | 32.9 (22.0)
  ALAT, Week 16, N=53, 53, 58, 56 | 25.7 (13.1) | 24.7 (14.4) | 24.3 (13.0) | 30.0 (25.3)

7. Secondary Outcome: Laboratory Safety Parameters (Biochemistry): Aspartate Aminotransferase (ASAT)
Description: Mean values at Week -4 and at Week 16
Time Frame: Week -4, Week 16
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | SIBA (D) | SIBA (E) | SIBA (D) M, W, F | IGlar
Number analyzed (Participants) | 57 | 59 | 62 | 61
IU/L
  ASAT, Week -4, N=56, 59, 62, 60 | 26.7 (13.6) | 22.5 (9.9) | 23.9 (8.5) | 24.2 (12.6)
  ASAT, Week 16, N=53, 53, 58, 56 | 23.3 (10.0) | 21.8 (7.7) | 21.7 (7.7) | 24.1 (13.7)

8. Secondary Outcome: Laboratory Safety Parameters (Biochemistry): Serum Creatinine
Description: Mean values at Week -4 and at Week 16
Time Frame: Week -4, Week 16
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | SIBA (D) | SIBA (E) | SIBA (D) M, W, F | IGlar
Number analyzed (Participants) | 57 | 59 | 62 | 61
umol/L
  Creatinine, Week -4, N=56, 59, 62, 60 | 74.5 (15.2) | 75.4 (19.0) | 73.2 (16.1) | 72.4 (13.9)
  Creatinine, Week 16, N=53, 53, 58, 56 | 76.1 (15.9) | 76.6 (19.1) | 71.5 (15.6) | 74.2 (14.4)

9. Secondary Outcome: Vital Signs: Diastolic Blood Pressure (BP)
Description: Mean values at baseline (Week 0) and at Week 16
Time Frame: Week 0, Week 16
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | SIBA (D) | SIBA (E) | SIBA (D) M, W, F | IGlar
Number analyzed (Participants) | 57 | 59 | 62 | 61
mmHg
  Week 0 (Baseline), N=57, 59, 62, 61 | 81 (9) | 82 (9) | 80 (8) | 79 (7)
  Week 16, N=55, 55, 60, 56 | 79 (8) | 82 (8) | 78 (9) | 77 (8)

10. Secondary Outcome: Vital Signs: Systolic Blood Pressure (BP)
Description: Mean values at baseline (Week 0) and at Week 16
Time Frame: Week 0, Week 16
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | SIBA (D) | SIBA (E) | SIBA (D) M, W, F | IGlar
Number analyzed (Participants) | 57 | 59 | 62 | 61
mmHg
  Week 0 (Baseline), N=57, 59, 62, 61 | 129 (14) | 131 (13) | 129 (15) | 127 (14)
  Week 16, N=55, 55, 60, 56 | 126 (14) | 131 (15) | 126 (16) | 128 (13)

11. Secondary Outcome: Vital Signs: Pulse
Description: Mean values at baseline (Week 0) and at Week 16
Time Frame: Week 0, Week 16
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | SIBA (D) | SIBA (E) | SIBA (D) M, W, F | IGlar
Number analyzed (Participants) | 57 | 59 | 62 | 61
beats/minute
  Week 0 (Baseline), N=57, 59, 62, 61 | 79 (10) | 79 (9) | 79 (9) | 76 (9)
  Week 16, N=55, 55, 60, 56 | 77 (11) | 78 (10) | 79 (9) | 74 (9)

12. Secondary Outcome: Physical Examination
Description: Physical examination was performed at screening (Week -4), randomisation (Week 0) and after 8 and 16 weeks of treatment. If any new findings or deterioration in previous findings were observed during the trial, these were recorded as AEs and are therefore not presented separately as no analysis was performed.
Time Frame: Week -4, Week 0, Week 8, Week 16
Arm/Group | SIBA (D) | SIBA (E) | SIBA (D) M, W, F | IGlar
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: The adverse events were collected in a time frame of 16 weeks + 5 days follow up
Description: Subjects in the safety analysis set contribute to the evaluation "as treated", hence the one subject who was treated with SIBA (D) 3W although he was randomised to SIBA (D) OD is analysed as SIBA (D) 3W for safety and as SIBA (D) OD in the FAS.
Arm/Group | SIBA (D) | SIBA (E) | SIBA (D) M, W, F | IGlar
Serious Adverse Events (participants affected / at risk) | 1/57 | 0/59 | 1/62 | 0/61
Other Adverse Events (participants affected / at risk) | 22/57 | 16/59 | 19/62 | 23/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SIBA (D) (N=57) | SIBA (E) (N=59) | SIBA (D) M, W, F (N=62) | IGlar (N=61)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SIBA (D) (N=57) | SIBA (E) (N=59) | SIBA (D) M, W, F (N=62) | IGlar (N=61)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 3 (3) | 3 (5) | 6 (7)
Toothache (Gastrointestinal disorders) | 3 (4) | 0 (0) | 2 (3) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 4 (4) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2) | 4 (4) | 7 (7)
Dyslipidaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 2 (2) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 5 (6) | 3 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 2 (4) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 3 (3) | 2 (2) | 5 (7) | 8 (9)
Paraesthesia (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 5 (6)
Hypertension (Vascular disorders) | 3 (3) | 1 (2) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.